CLINICAL TRIAL: NCT03657628
Title: Pilot Study of the Impact of a Physical Activity Intervention on Proliferation and Immune Markers in Benign Breast Tissue in Women With High Mammographic Breast Density
Brief Title: Physical Activity, Proliferation and Immune Markers in Benign Breast Tissue
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jennifer A. Ligibel, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 18-168; P50CA168504 (NIH)
Record Dates: First submitted 2018-08-24; First posted 2018-09-05 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical activity (Experimental): * The exercise intervention will consist of a supervised, moderate-intensity aerobic exercise program.
  * Will receive social/behavioral support
  * Will receive research staff contact time to encourage them to increase their physical activity level
  * The participants will be given the option of a third supervised session each week
  Interventions: Other: Exercise Intervention

INTERVENTIONS:
Other: Exercise Intervention — Strength training and moderate-intensity, aerobic exercise

SUMMARY:
This research study is evaluating the effect of exercise on markers in breast tissue and blood of premenopausal women who have been found to have dense breast tissue on mammogram.

DETAILED DESCRIPTION:
Women who exercise regularly have a lower risk of developing breast cancer, but the processes through which exercise could make cancer less likely to occur are not known. Some research in animals has shown that exercise can slow the growth of breast cancer cells and may increase the body's own defense mechanisms by stimulating the immune system. Very little is known about the effects of exercise on breast tissue in people. Understanding what changes occur in breast tissue and related markers in blood when a woman begins to exercise could provide more information about the ways in which exercise could prevent breast cancer.

The study is designed to look at the changes that occur in markers found in breast tissue and blood in women with dense breast tissue who take part in an exercise program. Density of breast tissue is a measure of how much of the breast tissue is made up of cells rather than fat. Breast density on mammogram has been linked to the risk of developing breast cancer, with women with higher degrees of breast density having a higher risk of developing breast cancer compared to women whose breasts are less dense.

Since the investigators do not know if these blood or breast tissue tests have any relationship to the development of breast cancer, the investigators do not plan to share the results of these tests with the participant or its physician. The investigators will give the participants the option of receiving the overall study results when the trial is completed, if the participant would like to receive them.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to any study-related procedures
* Premenopausal women, defined as:
* having regular menstrual cycles
* age ≤ 50 years with an intact IUD
* history of hysterectomy without oophorectomy
* Heterogeneously dense or very dense (BIRADS 3 or 4) breast tissue on mammogram within the last 3 years
* Physically inactive; engaging in <90 minutes of moderate or vigorous intensity PA per week
* No prior history of breast cancer
* At least 18 years old
* Physically able to exercise
* English speaking and able to read English

Exclusion Criteria:

* Self-reported inability to walk 2 blocks (at any pace)
* Prior history of breast cancer; prior DCIS is allowable as long as participant is not taking endocrine therapy and has at least 1 breast that has not been irradiated.
* On oral contraceptives; Mirena IUD is acceptable
* Cardiovascular, respiratory or musculoskeletal disease or joint problems that preclude moderate physical activity. Examples would include unstable angina, recent myocardial infarction, oxygen-dependent pulmonary disease, and osteoarthritis requiring imminent joint replacement. Moderate arthritis that does not preclude physical activity is not a reason for ineligibility.
* Psychiatric disorders or conditions that would preclude participation in the study intervention (e.g. untreated major depression or psychosis, substance abuse, severe personality disorder)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-09-17 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Impact of exercise upon expression of Ki-67 | 12-weeks
  To evaluate the change in breast tissue expression of Ki-67 in premenopausal women with increased breast density taking part in a 12-week physical activity intervention

SECONDARY OUTCOMES:
Changes in biomarker (IL-6) | 12-weeks
Changes in biomarker (TNF-a) | 12-weeks
Changes in biomarker (CRP) | 12-weeks
Changes in minutes of weekly physical activity | 12-weeks
  7-Day Physical Activity Recall Interview
Changes in waist to hip ratio | 12-weeks
Changes in weight (% change) | 12-weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Ligibel, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No